CLINICAL TRIAL: NCT04433793
Title: Yoga Intervention and Reminder E-mails for Reducing Cancer-related Fatigue - a Study Protocol of a Randomized Controlled Trial
Brief Title: Yoga Intervention for Reducing Fatigue in Cancer Patients
Acronym: Carfi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: German Cancer Aid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DRKS00016034
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Fatigue; Cancer
Keywords: Yoga; Mindfulness based Intervention; Fatigue; Cancer Patients
MeSH Terms: conditions — Fatigue; Neoplasms | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with cancer patients suffering from fatigue is planned. The study investigates the efficacy in terms of fatigue, depression and quality of life of eight-week yoga therapy (intervention group) compared to an 8-week waiting period without supportive intervention (control group).
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga group (Experimental): Patients in the yoga group will receive yoga therapy, one hour every week for eight weeks.
  Interventions: Behavioral: Yoga therapy
- Waitlist-control group (No Intervention): Patients in the waitlist-control group will receive no intervention at first, but nine weeks after IG, they will get the opportunity to also receive yoga therapy for 8 weeks.

INTERVENTIONS:
Behavioral: Yoga therapy — One yoga session will last one hour. It consists of physical exercises (asanas), conscious breathing (Pranayama) and deep relaxation (Savasana). The subsequent body exercises are structured from lying to sitting to standing. The following sequence of exercises will be repeated in each yoga unit: 1) Relaxation: conscious breathing, body scan, mindfulness 2) Vein pump 3) Pelvis and back rotation (adapted variation of the "nakrasana") 4) Pelvis opening (adapted variation of the "supta baddha konasana") 5) Shoulder bridge ("setu bandha sarvangasana) 6) Forward folds (Paschimottanasana and variations with Pranayama) 7) Backbend: intense east stretch (Purvottasana) 8) Diagonal static yoga cat (Majariasana 1 and resting pose) 9) Standing exercise 10) Upward Salute(Urdhva Hastasana) 11) Warrior 1 (Virabhadrasana 1) 12) Warrior 3 (Virabhadrasana 3) 13) Tree (Vrkasana variation) 14) Relaxation (Savasana).
  Arms: Yoga group

SUMMARY:
Cancer patients suffer from severe exhaustion and tiredness that is disproportionate to previous efforts and that cannot be completely reduced by sleep. The effectiveness of an 8 week yoga therapy (one hour a week) in patients with different cancer types on self-reported fatigue will be tested.

DETAILED DESCRIPTION:
Almost 90% of cancer patients suffer from symptoms of fatigue during treatment. Supporting treatments are increasingly used to alleviate the burden of fatigue. This study examines the short-term effects of yoga on fatigue, depression and quality of life. The aim of this study will evaluate the efficacy of yoga for cancer patients with mixed diagnoses reporting fatigue. We will randomly allocate 124 patients to an intervention group (N=62) receiving yoga and a wait-list control group (N=62) receiving yoga 9 weeks later. The yoga therapy will be performed in weekly sessions of 60 minutes each for 8 weeks. The primary outcome will be self-reported fatigue symptoms. Secondary outcome will be depression and Quality of life

ELIGIBILITY:
Inclusion Criteria:

* oncological disease
* planned to undergo cancer related treatment at radiotherapy outpatient clinic or the interdisciplinary oncological therapy outpatient clinic
* reported fatigue symptoms: (intensity ≥4, impairment ≥ 5).

Exclusion Criteria:

* insufficient knowledge of German
* severe emotional or physical impairment
* more than 50km distance to the university hospital which would require travelling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Changes from self-reported fatigue after participation in yoga therapy. | T0: At the beginning of the study, T1: after 9 weeks
  Self-reported cancer related fatigue; measured with: European Organisation for Research and Treatment of Cancer - Quality of life Questionnaire - Fatigue 13 (EORTC-QLQ-FA13); Scale 1-4; Higher scores mean a higher burden of fatigue

SECONDARY OUTCOMES:
Changes from Quality of life in cancer patients | T0: At the beginning of the study, T1: after 9 weeks
  self-reported Quality of life in cancer patients, measured with European Organisation for Research and Treatment of Cancer - Quality of life Questionnaire -Cancer 15 Palliativ (EORTC-QLQ-C15-Pal); Item 1- 14: Scale 1-4; Higher scores represent lower quality of life, Item 15: Scale 1-7; a higher value represents higher Overall Quality of life
Changes from Depression | T0: At the beginning of the study, T1: after 9 weeks
  self reported Depression, measured with patient health questionnaire -9 (PHQ-9); Scale: 1-4; higher score represents higher burden of depression

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Würzburg, Interdisciplinary Centre, Palliativ Medicine, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data that underlie results in publication (demographics and clinical characteristics, fatigue, Depression and Quality of life)
Supporting Information: Study Protocol, Analytic Code
Time Frame: starting 6 months after publication for 1 year
Access Criteria: for comparisons of efficacy of different yoga styles or supportive therapy in cancer patients

REFERENCES:
- [Background] Zetzl T, Schuler M, Renner A, Jentschke E, van Oorschot B. Yoga intervention and reminder e-mails for reducing cancer-related fatigue - a study protocol of a randomized controlled trial. BMC Psychol. 2019 Sep 18;7(1):64. doi: 10.1186/s40359-019-0339-3. PMID 31533823
- [Derived] Messer S, Oeser A, Wagner C, Wender A, Cryns N, Scherer RW, Mishra SI, Monsef I, Holtkamp U, Andreas M, Brockelmann PJ, Ernst M, Skoetz N. Yoga for fatigue in people with cancer. Cochrane Database Syst Rev. 2025 May 27;5(5):CD015520. doi: 10.1002/14651858.CD015520. PMID 40421669